CLINICAL TRIAL: NCT05083247
Title: Preoperative Treatment With mFOLFIRINOX (or Gem-Nab-P) +/- Isotoxic High-dose Stereotactic Body Radiation Therapy (iHD-SBRT) for Borderline Resectable Pancreatic Adenocarcinoma: a Randomised Phase II Study (STEREOPAC)
Brief Title: Preoperative mFOLFIRINOX (or Gem-Nab-P) +/- Isotoxic High-dose SBRT for Borderline Resectable Pancreatic Adenocarcinoma
Acronym: STEREOPAC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Collaborators: Jules Bordet Institute (Other); Belgian Group of Digestive Oncology (Other); University Hospital St Luc, Brussels (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ERA 001
Record Dates: First submitted 2021-09-29; First posted 2021-10-19 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-03

CONDITIONS: Pancreatic Neoplasm; Pancreatic Adenocarcinoma; Borderline Resectable Pancreatic Adenocarcinoma
Keywords: borderline resectable pancreatic cancer; neoadjuvant therapy; stereotactic body radiation therapy; chemotherapy
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: comparative randomised phase II
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Active Comparator): mFOLFIRINOX (oxaliplatin: 85 mg/m2, CPT-11: 165-180 mg/m2, folinic acid: 400mg/m2 and 5FU 2000-2400 mg/m2/46 h) regimen for 8 cycles every 2 weeks; or*Gemcitabine-Nab-P: gem: 1000 mg/m2 weekly 3 w/4; nab-P: 125 mg/m2 3 w/4 for 4 cycles in case of unfit for mFFX).
  Interventions: Drug: mFOLFIRINOX or Gemcitabine nab-paclitaxel; Procedure: Surgery
- Arm B (Experimental): mFOLFIRINOX for 6 cycles (or for 3 cycles Gemcitabine-Nab-P: gem: 1000 mg/m2 weekly 3 w/4; nab-P: 125 mg/m2 3 w/4 in case of unfit for mFFX) +Isotoxic high-dose SBRT: 5 x 7Gy with Simultaneous Integrated Boost (SIB) up to maximum 55Gy (= 1 week; starting ideally 2 weeks and maximum within 4 weeks after the end of chemotherapy)
  Interventions: Drug: mFOLFIRINOX or Gemcitabine nab-paclitaxel; Radiation: Isotoxic High-Dose (iHD)-SBRT; Procedure: Surgery

INTERVENTIONS:
Drug: mFOLFIRINOX or Gemcitabine nab-paclitaxel — oxaliplatin IV, irinotecan IV, leucovorin IV and 5-FU IV OR Gemcitabine IV Nab paclitaxel
  Other Names: mFFX or Gem/Nab-p
Radiation: Isotoxic High-Dose (iHD)-SBRT — Radiation therapy
  Arms: Arm B
Procedure: Surgery — Surgery

SUMMARY:
Surgical resection is the only potentially curative treatment for patients with pancreatic cancer with the aim of curative R0 resection and related improvement of survival. As a standard, surgery is usually followed by adjuvant therapy that improves survival but neoadjuvant therapy (NAT) is a rapidly emerging concept that needs to be explored and validated in terms of therapeutic options in borderline resectable pancreatic tumors. In this setting, preoperative FFX seems to be feasible and can be prolonged by radiation therapy. However, the exact and best therapeutic sequence is not yet known and the additional role of adding isotoxic high-dose stereotactic body radiotherapy (iHD-SBRT) to chemotherapy requires validation in randomised trials. We propose to evaluate the impact and efficacy of adding iHD-SBRT to preoperative neoadjuvant mFFX or Gem-NabP in patients with borderline resectable pancreatic adenocarcinoma.

DETAILED DESCRIPTION:
STEREOPAC is an multicenter, academic, prospective, randomised comparative, interventional study.

Patients receive 4 cycles of mFOLFIRINOX (or Gem-Nab-P)*. A full restaging (clinical, morphologic imaging, vascular involvement, biologics, CA 19.9) is performed. Non-progressive patients will be randomised (1:1) to

ARM A for receiving 4 additional cycles of chemo followed by surgery.

or to

ARM B for receiving 5th and 6th cycles of chemo then iHD-SBRT followed by a 7th (and optional 8th cycle) followed by surgery.

*: in case of CI or intolerance to mFFX, Gem-Nab-P regimen can be chosen or shifted to for 6 doses, then restaging, and then 3 doses followed by SBRT or 6 doses and immediate surgery)

Adjuvant chemotherapy administration is indicated unless the patient's condition precludes it.

ELIGIBILITY:
Inclusion criteria:

* Cytologic or histologic proof of adenocarcinoma of the pancreatic head or uncinated process or body or tail. Diagnosis should be verified by local pathologist
* cTNM stage: T1-4N0-2M0
* Confirmation of clinical and radiographic stage as borderline resectable (CT scan and/or MRI scan with contrast according to the NCCN criteria) by a multidisciplinary board, composed by a dedicated oncological surgeon, radiologist and GI oncologist)
* Age > 18 years old
* No prior chemotherapy or radiation for pancreatic cancer
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* No grade ≥ 2 neuropathy
* Laboratory parameters as follows:
* Absolute neutrophil count (ANC) ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 9 g/dL
* Creatinine ≤ 1.5 x upper limit of normal (ULN) or estimated GFR >45 mL/min
* Bilirubin ≤ 1.5 x ULN, including after adequate biliary stenting with metal stent (ideally 4 cm length)
* Aspartate aminotransferase (AST) / alanine aminotransferase (ALT) ≤ 2.5x ULN
* CA 19.9 < 2500 kU/l (baseline, prior to any therapy and absence of cholestasis)

Exclusion Criteria:

* Evidence of extrapancreatic disease on diagnostic imaging (CT, MRI or PET scan), histologically proven or at laparoscopy, including distal nodal involvement beyond the peripancreatic tissues (including non-regional lymph node involvement, ie: proven involvement of precaval lumbar lymphadenopathy(ies) and/or distant metastases
* Locally advanced disease as defined by the NCCN criteria (version 2.2021) ie > 180° arterial encasement (SMA and CA) unreconstructible venous encasement (SMV/PV) due to tumor involvement or occlusion of a long segment.
* CA 19.9 > 2500 kU/l (baseline and absence of cholestasis)
* Contraindication of surgery (general)
* Contraindications to receive FFX or gemcitabine-nab-Paclitaxel
* History of radiotherapy of the upper abdomen
* Prior treatment with oxaliplatin, irinotecan, fluoruouracil or capecitabin
* Patient < 18 years old
* Major surgery within 4 weeks of study entry
* Uncontrolled pre-existing disease including, but not limited to: active infection, symptomatic congestive heart failure, unstable angina, social / psychiatric disorder that would limit compliance to treatment and good understanding of the informed consent form
* Other concurrent anticancer therapies
* Existence of another active neoplasia other than basal cell carcinoma of the skin, cervical carcinoma in situ or non-metastatic prostate cancer. Patients who have a history of neoplasia must have been in remission for more than 5 years to be included in the protocol
* Pregnant or breastfeeding women; for women of childbearing potential only, a negative pregnancy test done < 7 days prior to registration is required. Using of reliable contraception for at least 1 month before treatment is mandatory
* Chronic concomitant treatment with strong inhibitors of cytochrome p450, family 3, subfamily a, polypeptide 4 gene (CYP3A4) is not allowed on this study; patients on strong CYP3A4 inhibitors must discontinue the drug for 14 days prior to registration on the study

Additional exclusion criteria before randomisation:

* Progressive disease (RECIST or PETCT, including non locoregional nodal involvement and increase of CA 19.9 by 20%) after receiving 4 cycles of FFX (or G/NP), including shift chemotherapy in case of early progression.
* CA 19.9 > 1000 kU/l after neoadjuvant therapy.
* Presence of unmanageable toxicity during the first part of neoadjuvant chemotherapy (first 4 cycles or 6 doses of FFX or G/NP, respectively.
* Pancreatic tumour > 7.0 cm in greatest axial dimension at the time of randomization
* Massive invasion of the stomach or intestines and/or direct intestinal invasion of the mucosae visible at ultrasoundendoscopy
* Active gastric or duodenal ulcer disease at the time of randomization. Tolerated in case of antecedent without active ulcer (confirmation by endoscopy before iHD-SBRT)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2023-03-24 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 weeks
  Defined as time from randomisation to the first documentation of event where events considered are 1) disease progression, per RECIST, prior to surgery, 2) discovery of hepatic or peritoneal carcinomatosis during surgical exploration, 3) recurrent disease following R0-R1 surgery, or 4) death due to any cause.
R0 Resection rate | up to 12 months
  Defined as the proportion of eligible randomised patients in whom a R0 resection was achieved during surgery after neoadjuvant treatment with FOLFIRINOX +/- iHD-SBRT. R0 resection indicates a microscopically margin-negative resection (>1 mm) from the inked margins (pancreatic transection, vascular and posterior circumferential resection margins).

SECONDARY OUTCOMES:
Resection rate | up to 12 months
  defined as the percentage of eligible randomised patients that underwent a curative-intent resection
Pathologic complete/major response (pCR) | up to 12 months
  Defined as the proportion of patients in whom a pCR or a major (<10% of residual tumour cells) was confirmed by histopathologic review of the surgical specimen.
Complete feasibility of the therapeutic sequence | up to 12 months
  Defined as the proportion of patient who performed completely the neoadjuvant therapeutic sequence with mFFX (or Gem-Nab-P) +/- iHD-SBRT until surgery (abdominal exploration with or without pancreatectomy). The therapeutic sequence will not be considered as feasible if less than 60% of patients do not complete it until surgery.
Overall survival (OS) | Defined as the time interval between randomisation and death, assessed up to 60 months
  Defined as the time interval between randomisation and death. 95% confidence interval will be estimated based on standard method.
Locoregional failure free interval (LFFI) | defined as the time interval between the randomisation and the 1st documented date of locoregional failure, assessed up to 60 months
  defined as the time interval between the randomisation and the date of locoregional failure. A locoregional failure is any progressive or recurrent pancreatic cancer in the original tumour location or the N1-2 lymph node areas
Distant metastases free interval (DMFI) | defined as the period of time without distant metastasis after randomisation, assessed up to 60 months
  defined as the period of time without distant metastasis after randomisation.
Toxicity, Incidence of adverse events | up to 24 months
  assessed per Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 and the Patient-Reported Outcomes version of the CTCAE
Postoperative complications | up to 12 months
  defined according to the Clavien-Dindo classification and definitions of post-pancreatic surgery complications (pancreatic fistula, delayed gastric emptying and bleeding) by the International study group on Pancreatic Surgery.
Quality of life (QoL) assessment - General | up to 24 months
  assessed per EORTC General Quality of life of Cancer patient questionnaire QLQ-C30 version 3.0 (minimum value: 30 - maximum value: 126; higher score associated with worse QoL outcome).
Quality of life (QoL) assessment - Pancreatic cancer | up to 24 months
  assessed per EORTC Quality of life of Pancreatic Cancer patient questionnaire QLQ-PAN26 (minimum value: 26 - maximum value: 104; higher score associated with worse QoL outcome).
Quality of life (QoL) assessment - Depression | up to 24 months
  assessed per the depression test : Patient Health Questionnaire-9 (PHQ-9; minimum value: 0 - maximum value: 27; higher score associated with worse QoL outcome)
Technical and quality success rate of EUS-delivered fiducials. | up to 12 months
  The technical success is defined as at least one marker presumed to be inside the tumour at the end of the EUS procedure. The quality success is defined as a score equal or higher than 6/12 points based on the 5 items quality score defined in [Figueiredo M, Bouchart C et al 2021].

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc Van Laethem, MD, Study Chair — Erasme Hospital, ULB; Christelle Bouchart, MD, Principal Investigator — Jules Bordet Institute
Locations (10):
- Belgium (10):
  - Uza Antwerp, Antwerp
  - Hopital Erasme, HUB, Brussels
  - Jules Bordet Institute, HUB, Brussels
  - CHIREC, Brussels
  - Cliniques Universitaires St luc, Brussels
  - UZ Gent, Ghent
  - AZ Groeninge, Kortrijk
  - Pôle Hospitalier Jolimont, La Louvière
  - Clinique Chc Montlégia, Liège
  - CHU Ambroise Paré, Mons

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Figueiredo M, Bouchart C, Moretti L, Mans L, Engelholm JL, Bali MA, Van Laethem JL, Eisendrath P. EUS-guided placement of fiducial markers for stereotactic body radiation therapy in pancreatic cancer: feasibility, security and a new quality score. Endosc Int Open. 2021 Feb;9(2):E253-E257. doi: 10.1055/a-1324-2892. Epub 2021 Feb 3. PMID 33553589
- [Background] Bouchart C, Engelholm JL, Closset J, Navez J, Loi P, Gokburun Y, De Grez T, Mans L, Hendlisz A, Bali MA, Eisendrath P, Van Gestel D, Hein M, Moretti L, Van Laethem JL. Isotoxic high-dose stereotactic body radiotherapy integrated in a total multimodal neoadjuvant strategy for the treatment of localized pancreatic ductal adenocarcinoma. Ther Adv Med Oncol. 2021 Oct 19;13:17588359211045860. doi: 10.1177/17588359211045860. eCollection 2021. PMID 34691244
- [Background] Manderlier M, Navez J, Hein M, Engelholm JL, Closset J, Bali MA, Van Gestel D, Moretti L, Van Laethem JL, Bouchart C. Isotoxic High-Dose Stereotactic Body Radiotherapy (iHD-SBRT) Versus Conventional Chemoradiotherapy for Localized Pancreatic Cancer: A Single Cancer Center Evaluation. Cancers (Basel). 2022 Nov 22;14(23):5730. doi: 10.3390/cancers14235730. PMID 36497212
- [Derived] Bouchart C, Navez J, Borbath I, Geboes K, Vandamme T, Closset J, Moretti L, Demetter P, Paesmans M, Van Laethem JL. Preoperative treatment with mFOLFIRINOX or Gemcitabine/Nab-paclitaxel +/- isotoxic high-dose stereotactic body Radiation Therapy (iHD-SBRT) for borderline resectable pancreatic adenocarcinoma (the STEREOPAC trial): study protocol for a randomised comparative multicenter phase II trial. BMC Cancer. 2023 Sep 21;23(1):891. doi: 10.1186/s12885-023-11327-x. PMID 37735634